CLINICAL TRIAL: NCT01157598
Title: Efficacy of Bispectral Index Monitoring for Midazolam and Meperidine Induced Sedation During Endoscopic Submucosal Dissection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Samsung Medical Center IRB, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2009-08-037
Record Dates: First submitted 2010-07-05; First posted 2010-07-07 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Gastric Adenoma; Gastric Cancer
Keywords: gastric adenoma; early gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- BIS group (Active Comparator)
  Interventions: Device: bispectral index monitoring
- non BIS group (Placebo Comparator)
  Interventions: Device: bispectral index monitoring

INTERVENTIONS:
Device: bispectral index monitoring — parameter monitoring of bispectral index

SUMMARY:
Background: Endoscopic submucosal dissection (ESD) usually requires adequate level of sedation due to lengthy and uncomfortable procedure. Propofol induced sedation with bispectral index (BIS) monitoring has been reported to lead to higher satisfaction of patients and endoscopists during ESD. However, there is no data about efficacy of midazolam and meperidine induced sedation with BIS monitoring during ESD. This study was to evaluate whether midazolam and meperidine induced sedation with BIS monitoring could improve the satisfaction and reduce the dose of midazolam and meperidine during ESD.

ELIGIBILITY:
Inclusion Criteria:

* gastric adenomas, differentiated-type gastric cancers greater than 30 mm in diameter without ulceration and gastric cancers up to 30 mm with ulceration, or minute submucosal invasion

Exclusion Criteria:

* if they were under 18 years of age
* had an ASA classification of 4-5
* were pregnant
* had a history of stroke or an allergy to sedative drugs.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
the satisfaction of patients and endoscopist in midazolam and meperidine induced sedation with BIS monitoring during ESD | within the one day after ESD

SECONDARY OUTCOMES:
the dose of midazolam and meperidine during ESD with BIS monitoring | within one hour after ESD

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea